CLINICAL TRIAL: NCT06685614
Title: Orthodontic Bracket Bonding (OBB)
Brief Title: Orthodontic Bracket Bonding
Acronym: OBB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202405087RIND
Record Dates: First submitted 2024-11-03; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Bracket Bonding
Keywords: computer-aided design and computer-aided manufacturing; orthodontics; bracket bonding; digital dentistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- direct (Active Comparator): traditional direct bonding
  Interventions: Device: orthodontic bracket bonding
- indirect (Active Comparator): traditional indirect bonding, bracket transfer tray made using cast model
  Interventions: Device: orthodontic bracket bonding
- 3D-printed tray (Experimental): virtual bracket bonding and 3D print out indirect bracket bonding transfer tray using CAD/CAM technique
  Interventions: Device: orthodontic bracket bonding
- 3D-printed model (Experimental): virtual bracket bonding and 3D print out digital model with brackets; indirect bracket bonding transfer tray made using 3D-printed model
  Interventions: Device: orthodontic bracket bonding

INTERVENTIONS:
Device: orthodontic bracket bonding — compare the effectiveness of different bonding methods including traditional direct bonding, traditional indirect bonding, indirect bonding using 3D-printed transfer tray, and indirect bonding using vacuum-formed transfer tray made with 3D-printed models

SUMMARY:
Accurate bracket positioning is crucial for effective fixed orthodontic treatment and a core component of orthodontic specialist training. Clinically, two main bonding techniques exist: direct and indirect. Due to limited high-quality trials, there is no conclusive evidence favoring direct or traditional indirect bonding for accuracy. Advances in digital dentistry have further optimized indirect bonding; 3D software allows orthodontists to position virtual brackets for digital tooth alignment, and CAD/CAM technology enables the production of digitally assisted transfer trays. This project will conduct a prospective randomized controlled trial to compare the effectiveness of different bonding methods including traditional direct bonding, traditional indirect bonding, indirect bonding using 3D-printed transfer tray, and indirect bonding using vacuum-formed transfer tray made with 3D-printed models. Outcomes will include bracket placement accuracy, chairside time, bonding failure rate, treatment adjustments, and cast-radiograph evaluation. Despite current costs of CAD/CAM in orthodontics, this study aims to train orthodontic residents, optimize patient care, and foster collaboration across orthodontic specialists and industry. The alternative hypotheses are: (1) Significant differences exist in bracket positioning accuracy across bonding techniques; (2) Bonding techniques vary significantly in chairside time, bonding failure rates, incidence of bracket repositioning, and additional tooth adjustments.

DETAILED DESCRIPTION:
Participants for this study will be recruited from the Department of Orthodontics at National Taiwan University Hospital (NTUH). Given that younger children may have incomplete tooth eruption, short clinical crowns, and challenges with behavioral control, this study will include only patients aged 20 and older. Eligible participants will be those undergoing comprehensive, non-extraction orthodontic treatment with complete dentition (excluding wisdom teeth) and thorough documentation, including panoramic and lateral cephalometric radiographs, models, and intraoral scans. For eligible patients, informed consent will be obtained prior to treatment, and they will be randomized into different groups to receive bracket bonding using various techniques according to the randomization protocol. Random assignment will be block-stratified and conducted with assistance from an independent statistician, with expert oversight ensuring all patients are correctly allocated.

All first-year orthodontic residents at NTUH will participate in this study as bracket positioning is a fundamental component of their orthodontic training. These residents will receive lectures on traditional direct bonding procedures and hands-on training in digital orthodontic techniques, supported by standard operating procedure manuals for each bonding technique. As all procedures align with standard clinical practice, no additional patient risks or protective measures are needed.

For patients who have undergone virtual bonding before actual bonding, an intraoral scan will be taken post-bonding to assess differences between planned and actual bracket placement. All participants will adhere to a treatment schedule with appointments every three to four weeks, advancing according to the supervising orthodontist's evaluations. Upon treatment completion, documentation will include panoramic and lateral cephalometric radiographs, impressions, intraoral scans, and retainer fabrication.

Statistical analysis will be conducted using SPSS (Version 20; IBM Corp., Armonk, NY, USA). The study will assess the accuracy of bracket placement and evaluate correlations between pre-treatment occlusion and post-treatment outcomes across different bonding techniques.

ELIGIBILITY:
Inclusion Criteria:

i. Patients with a fully erupted permanent dentition. ii. Orthodontic treatment plans that do not require extractions (excluding wisdom teeth).

iii. Patients who have not previously undergone orthodontic treatment. iv. Complete dentition (excluding wisdom teeth). v. Adult patients aged 20 years or older.

Exclusion Criteria:

i. Patients requiring extraction of teeth other than wisdom teeth. ii. Fixed prostheses on teeth other than molars. iii. Significant tooth morphology defects requiring fixed prosthetic restorations.

iv. Missing teeth (excluding wisdom teeth). v. Patients with fractured crowns or large restorations on the buccal surfaces of crowns.

vi. Teeth with severe rotation or crowding that may impede direct bonding or tray placement.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2029-11-09 (Estimated); Study Completion 2029-11-09 (Estimated)

PRIMARY OUTCOMES:
treatment outcomes | Post-treatment: completion of orthodontic treatment, at time of bracket debonding
  cast-radiograph evaluation (according to the grading system for dental casts and panoramic radiographs by the American Board of Orthodontics)

SECONDARY OUTCOMES:
accuracy of bracket placement | Immediate after bracket bonding
  accuracy of bracket placement compared to virtual bonding (using 3D superimposition of the digital models)

IPD SHARING:
Plan to Share IPD: No